CLINICAL TRIAL: NCT02556762
Title: Phase III Randomized Controlled Trial of Definite Chemoradiotherapy in Patients With Esophageal Cancer: Simultaneous Modulated Accelerated Boost Versus Standard Dose Radiotherapy
Brief Title: Simultaneous Modulated Accelerated Boost Versus Standard Dose Radiotherapy in Esophageal Cancer
Acronym: SUMC-EC-002
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chuangzhen Chen (Other)
Responsible Party: Sponsor-Investigator, Chuangzhen Chen, M.D, Shantou University Medical College
Organization: Shantou University Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUMC-EC-002
Record Dates: First submitted 2015-09-17; First posted 2015-09-22 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; Simultaneous modulated accelerated boost; Standard dose radiotherapy; Chemotherapy; Survival
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMART boost (Experimental): Radiotherapy with simultaneous modulated accelerated boost
  Interventions: Radiation: Radiotherapy with simultaneous modulated accelerated boost; Drug: PF
- Standard dose RT (Active Comparator): Standard dose radiotherapy
  Interventions: Radiation: Standard dose radiotherapy; Drug: PF

INTERVENTIONS:
Radiation: Radiotherapy with simultaneous modulated accelerated boost — Radiotherapy: 66Gy/30F to the gross tumor and 50Gy/25 to subclinical diseases
  Other Names: SIB
  Arms: SMART boost
Radiation: Standard dose radiotherapy — Radiotherapy: 50Gy/25F to both gross tumor and subclinical disease
  Arms: Standard dose RT
Drug: PF — Chemotherapy: Cisplatin and 5fluorouracil

SUMMARY:
This randomized phase III trial is to compare simultaneous modulated accelerated boost with standard dose radiotherapy given together with chemotherapy in treating patients with esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of primary squamous cell carcinoma of the esophagus.
* Primary disease at cervical, upper or middle thoracic esophagus
* T1-4, N any, M0 (except supraclavicular lymph node).
* Age≥18 & ≤75.
* ECOG score 0-2.
* Platelets ≥ 150,000, Hgb ≥ 10 gm%, ANC ≥ 1500, serum creatinine ≤ 1.5 mg/dl.
* Adequate liver function.
* Patients with prior malignancy are eligible if disease-free ≥ 5 years.
* No prior chest radiotherapy, systemic chemotherapy or major esophageal surgery.
* Signed study-specific informed consent form prior to study entry.

Exclusion Criteria:

* Patients with tracheo-esophageal fistula.
* Patients with invasion into mucosa of trachea or major bronchi.
* Patients with uncontrolled serious medical or mental illnesses.
* Prior RT that would result in overlap of planned RT fields.
* Pregnancy or women of childbearing potential and men who are sexually active
* Women who are breastfeeding a baby.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2015-08; Primary Completion 2022-03-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years

SECONDARY OUTCOMES:
Local-regional control | 2 years
Distant metastasis-free survival | 2 years
Disease-free survival | 2 years after randomization
Acute and late toxicities using CTCAE v4.0 | 2 years
  The probabilities of grade ≥ 3 acute toxicities and 2-year late toxicities of esophagus and lungs.
Quality of life as assessed with FACT-E | 2 years
  FACT-E score
Quality of life as measured with EQ-5D | 2 years
  The score of EQ-5D questionnaire
Biomarkers | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chuangzhen Chen, MD, Principal Investigator — Cancer Hospital, Shantou University Medical College
Locations (1):
- Cancer Hospital, Shantou University Medical College, Shantou, Guangdong, China